CLINICAL TRIAL: NCT04500795
Title: Prospective Study on the Use of Middle Meningeal Artery Embolization for Chronic Subdural Haematoma
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Update in other trial results
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, George KC Wong, Professor, Chinese University of Hong Kong
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GWMMAE01
Record Dates: First submitted 2020-08-04; First posted 2020-08-05 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Chronic Subdural Hematoma; Subdural Hematoma
Keywords: chronic subdural hematoma; subdural hematoma; head injury; middle meningeal artery; hemorrhage; embolization
MeSH Terms: conditions — Hematoma, Subdural, Chronic; Hematoma, Subdural; Craniocerebral Trauma; Hemorrhage

STUDY DESIGN:
Intervention Model Description: Patients divided into two groups, embolization group and control (conventional) group. Patients remain in control group if they refuse embolization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Embolization Group (Experimental): Patients with residual or recurrent haematoma (higher than 10mm thickness of haematoma at any dimension) following prior surgical evacuation of haematoma will be admitted to the Embolization Group and undergo embolization of MMA. Serial CT scans will be taken at times of presentation of the residual or recurrent haematoma, 1-day, 1-week, 1-month, 3-month, and 6-month following embolization. Size of haematoma will be measured for comparison to the Control Group. Clinical examinations will be done at the same setting.
  Interventions: Procedure: Middle meningeal artery embolization
- Control Group (No Intervention): All symptomatic patients (headache unresponsive to analgesic or neurological deficits including focal neurological deficits, deteriorated consciousness, headache, seizures, and other signs or symptoms suggestive of SDH as the cause) will undergo haematoma evacuation either by burr-hole drainage or craniotomy. Their response to treatment, neurological status, and CT scans will be monitored. Asymptomatic patients will be monitored radiologically (CT) every 2-4 weeks. The decision for surgical evacuation of haematoma will be based on CT findings (increasing haematoma size) and presentation of symptoms or neurological deficits. They remain in the control group should they refuse embolization of MMA. The size of haematoma will be measured continuously based on CT scans taken at times of presentation, 1-day, 1-week, 1-month, 3-month, and 6-month post-op. Size of haematoma, residual or recurrent will be measured for comparison to the Embolization Group.

INTERVENTIONS:
Procedure: Middle meningeal artery embolization — MMA embolization will be performed with a liquid embolization agent with local anaesthesia. Selective angiography will be performed before embolization to select MMA branch targets and detect potentially dangerous collateral vessels. If no dangerous collaterals are found, MMA branches supplying to the dura of convexity will be targeted and embolized according to findings of the selective angiography using a liquid embolization agent. If dangerous collaterals are identified, the microcatheter will be advanced more distally or the collaterals will be coiled prior to embolization. Procedure will be concluded once the flow stasis of MMA is confirmed. Embolization is considered successful if all MMA targets are embolized without procedural complications.
  Patients with existing use of antiplatelet or anticoagulation medication will not undergo medication reversal for the embolization procedure.
  Arms: Embolization Group

SUMMARY:
Subdural haematoma is a common neurosurgical condition that results in different levels of neurological deficits in patients. It can be further classified into acute and chronic, which have different pathophysiology. Acute haematoma is a common result of traumatic injuries involving the tearing of the bridging veins, while chronic subdural haematoma can be both a result of traumatic injuries or recurrence following surgical management of the acute counterpart. For symptomatic patients, they are often surgically managed by haematoma drainage via burr-hole drainage and craniotomy. Recurrent bleeding following close monitor or surgical evacuation of haematoma is however very high. Recent studies approximate the recurrence rate of 2%-33.3%. Recent evidence suggests the angiogenesis of middle meningeal arteries (MMA) in response to inflammation and healing process contributes to the development of chronic subdural haematoma, and its high recurrence chance. Several studies have looked into the use of middle meningeal artery embolization to halt the bleeding of a chronic subdural haematoma, and have found promising results in terms of haematoma reduction and prevention of surgical rescues.

DETAILED DESCRIPTION:
The primary goal of the study is to assess the safety and efficacy of middle meningeal artery embolization in treating patients presenting with subdural haematoma. Previous studies and trial in other countries have shown promising results. This study aims to serve as the pilot clinical study of the procedure in Hong Kong and setting the ground work for a future multi-centre randomised trial.

Patients presenting with subdural haematoma will be assessed clinically and radiologically. Patients' demographic information, clinical information, and past medical history will be recorded for the purpose of the study. Symptomatic patients will undergo haematoma removal either by burr-hole drainage or craniotomy. They will undergo a series of CT-scans before and after treatment to assess the characteristics of the haematoma (size, side, site, composition of the haematoma, etc). Patients will then be divided into the embolization group and the control group. Patients with residual or recurrent haematoma (higher than 10mm thickness of haematoma at any dimension) following prior surgical evacuation of haematoma will be admitted to the Embolization Group and undergo embolization of MMA. Serial CT scans will be taken at times of presentation of the residual or recurrent haematoma, 1-day, 1-week, 1-month, 3-month, and 6-month following embolization. Size of haematoma will be measured for comparison to the Control Group. Clinical examinations will be done at the same setting. For the control group, after the initial treatment of haematoma removal, they will be monitored clinically for signs of neurological deficits, presentation of symptoms. They remain in control group should they refuse entering the MMA embolization group. They will have the same clinical and radiological follow-up as the embolization group.

MMA embolization will be performed with a liquid embolization agent with local anaesthesia. Selective angiography will be performed before embolization to select MMA branch targets and detect potentially dangerous collateral vessels. If no dangerous collaterals are found, MMA branches supplying to the dura of convexity will be targeted and embolized according to findings of the selective angiography using a liquid embolization agent. If dangerous collaterals are identified, the microcatheter will be advanced more distally or the collaterals will be coiled prior to embolization. Procedure will be concluded once the flow stasis of MMA is confirmed. Embolization is considered successful if all MMA targets are embolized without procedural complications.

Patients with existing use of antiplatelet or anticoagulation medication will not undergo medication reversal for the embolization procedure.

Patients will be discharged following treatment based on the results of the post-operative assessments.

ELIGIBILITY:
Inclusion Criteria:

* Patients (age 18 or above) with chronic subdural haematoma diagnosed by computed tomography and clinical presentation.

Exclusion Criteria:

* SDH with thickness of 10mm or less, lack of mass effect.
* SDH secondary to existing conditions (brain tumour, arachnoid cyst, spontaneous intracranial hypotension, previous craniotomy not due to chronic SDH)
* Patients in poor medication condition or with life expectancy less than 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Percentage volume change of recurrent haematoma | From date of recruitmnent until the date of first documented progression or date of death from any cause or at 6 months, whichever came first
  Primary outcome of the studies is the percentage volume change of recurrent haematoma measured by serial CT brain scans after embolization (embolization group) or haematoma removal (control group).

SECONDARY OUTCOMES:
Number of patients with treatment failure | From date of recruitment until the date of first documented progression or date of death from any cause or at 6 months, whichever came first
  Secondary outcome is number of patients with treatment failure. Treatment failure is defined as Patients presenting with reaccumulating or residual haematoma (haematoma thickness >10mm) following embolization or haematoma removal by the sixth month of follow-up; or patients requiring surgical rescue due to the recurrence of haematoma or surgical or endovascular complications.
Number of patients with 30-day morbidities and mortality | 30 days following the day of recruitment
  Number of patients with 30-day morbidities and mortality. 30-day morbidities include adverse events of different severity. Severe adverse events (excluding death) include prolonged intubation longer than 48 hours, return to OR, unplanned reintubation, deep vein thrombosis or pulmonary embolism, coma, sepsis or septic shock, stroke, myocardial infarction, surgical site or deep infection, acute renal failure. Minor adverse events include urinary tract infection, pneumonia, progressive renal insufficiency, and neurological deficits (residual or new).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery, The Chinese University of Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: Undecided
Not decided yet.